CLINICAL TRIAL: NCT01012830
Title: Huperzine-A for Cognitive Dysfunction and Functional Status in Schizophrenia
Brief Title: Huperzine-A to Help With Mental Problems and the Inability to Care for Onself in Patients With Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Collaborators: American Legion of Iowa Foundation (Other)
Responsible Party: Prasad R. Padala, M.D., VA Nebraska Western Iowa Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 636-631
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Schizophrenia; Dementia
Keywords: Schizophrenia; Cognitive Disorders; Dementia; Huperzine A; HupA
MeSH Terms: conditions — Schizophrenia; Dementia; Cognitive Dysfunction | interventions — huperzine A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Huperzine A (Experimental): 200 micrograms (mcg) of HuperzineA taken twice daily.
  Interventions: Drug: Huperzine A

INTERVENTIONS:
Drug: Huperzine A — Huperzine A in 200 microgram (mcg) capsules taken twice daily for 8 weeks.
  Other Names: HupA; Huperzine-A; Huperzia serrata

SUMMARY:
Use Huperzine-A, a herbal supplement normally used for treatment of Alzheimer's disease, to potentially improve cognitive dysfunction (memory problems) and functional capacity (ability to perform common daily tasks such as cooking, bathing, telephone, shopping) in people with schizophrenia.

DETAILED DESCRIPTION:
HupA, an alkaloid initially identified from the Chinese herbal medicine Huperia serrata, is a potent reversible acetyl cholinesterase (AChE) inhibitor with additional unique properties including NMDA-receptor antagonist properties, neuroprotective and antioxidant effects. In animal studies, HupA was shown to possess greater inhibitory, longer-lasting, and more selective effects on AChE activity than donepezil. In clinical studies HupA improved memory, mood, and activities of daily living in patients with Alzheimer's dementia. Adverse effects have been reported at a very low rate in all the clinical trials, and are mainly cholinergic, such as dizziness, nausea, gastrointestinal symptoms, headaches and depressed heart rate. Thus, HupA is an attractive option which may have beneficial effects not only on cognitive but also functional domains of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. age 19-59
2. diagnosis of schizophrenia by MINI
3. cognition score 1 standard deviation below published norms in controls
4. clinically stable for 12 weeks i.e. on the same antipsychotic(s) for 8 weeks and stable dose for at least 4 weeks
5. have no more than moderate severity rating on hallucinations, delusions formal thought disorder (BPRS), negative symptoms (PANSS_N)
6. minimal EPS (Simpson-Angus <6)
7. minimal depression (Calgary <10)
8. stable dose of other psychotropics (2 months)
9. not pregnant.

Exclusion Criteria:

1. history of active peptic ulcer disease within 1 year of screening
2. clinically significant cardiac arrhythmia
3. resting pulse less than 50
4. active cancer (skin tumors other than melanoma are not excluded)
5. history of clinically significant stroke
6. current evidence or history in the past 2 years of epilepsy, focal brain lesion
7. start of cholinesterase inhibitors/ cognitive enhancers (galantamine, rivastigmine, donepezil, vitamin E and memantine) within 2 months of screening, 8. use of medications with significant central nervous system anticholinergic activity within 2 months of screening.

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery | First visit, 4 weeks, 8 weeks

SECONDARY OUTCOMES:
University of California Performance Skills Assessment-Brief (UPSA-B) | First visit, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prasad R Padala, MD, MS, Principal Investigator — VA Office of Research and Development
Locations (1):
- Veterans Affairs Nebraska Western Iowa Health Care System, Omaha, Nebraska, United States